CLINICAL TRIAL: NCT03318159
Title: Open Label, Phase II Study Investigating the Efficacy of Posaconazole as Prophylaxis Antifungal Agent in Aplastic Anemia / Hypoplastic Myelodysplastic Syndrome Patients Undergoing Antithymocyte Globulin Treatment
Brief Title: Posaconazole Prophylaxis During ATG Treatment for hMDS/AA Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, YOUNGIL KOH, assistant professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-1706-207-866
Record Dates: First submitted 2017-10-10; First posted 2017-10-23 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Aplastic Anemia; Myelodysplastic Syndromes; Fungal Infection
MeSH Terms: conditions — Anemia, Aplastic; Myelodysplastic Syndromes; Mycoses | interventions — posaconazole

STUDY DESIGN:
Intervention Model Description: open label, single arm, phase 2, multicenter
  *historical control will be used for comparison: historical control patients are defined as those diagnosed with AA/hMDS and underwent ATG treatment with either fluconazole or itraconazole prophylaxis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- posaconazole prophylaxis group (Other): aplastic anemia / hypoplastic myelodysplastic syndrome patients undergoing antithymocyte globulin treatment and receiving posaconazole as prophylaxis antifungal agent
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Posaconazole — Dosing of posaconazole Posaconazole tablet 300 mg twice daily on day 1; Maintenance dose: 300 mg once daily on day 2 and thereafter. Treatment period: 4 weeks
  *if posaconazole tablet intolerance: posaconazole suspension 200mg tid

SUMMARY:
To investigate the efficacy of posaconazole as prophylaxis antifungal agent in aplastic anemia / hypoplastic myelodysplastic syndrome (AA/hMDS) patients undergoing antithymocyte globulin (ATG) treatment

DETAILED DESCRIPTION:
With compromised bone marrow function, patients with aplastic anemia (AA) and/and hypoplastic myelodysplastic syndrome (hMDS) are at an increased risk of invasive fungal infection. Moreover, the use of antithyocyte globulin (ATG), a part of standard first line treatment for AA/hMDS, increases the risk of fungal infection due to its antilymophocytic effects. It has been reported that fungal infection occurs most often in the first few weeks after initiation of ATG treatment, and the reported incidence of fungal infection overall varies from 9~80% for AA/hMDS patients. Among them invasive fungal infection accounts for 6-20% depending on reports. Such being the case, antifungal prophylaxis is recommended for AA/hMDS patients undergoing ATG treatment. More specifically, the British Committee for Standards in Haematology (BCSH) recognized the threat of increased invasive fungal infections in AA patients, and stipulated the use of mould (aspergillus) active azole, "preferably itraconazole or posaconazole" as prophylaxis. Unfortunately however, though many centers have adopted their own practice schemes, and antifungals have been routinely administered in the context of investigational regimens, there is no consensus as to which antifungal agent should be used.

Considering Aspergillus sp has remained the most common fungal isolate in AA patients for the past 20 years, it is only rational that an antifungal agent with broad spectrum, covering both yeast and fungi, be used in this context. Posaconazole, a triazole antifungal agent, not only has a broad coverage spectrum but also associated with predictable and reliable systemic bioavailability. Also for patients, once daily dosage is both pragmatic and convenient. According to meta-analyses of prophylactic antifungal agents use (published in 2007), fluconazole diminished the risk of fungal related mortality compared to placebo (RR 0.49, 95% CI: 0.32-0.75, P=0.0009). More importantly, when compared to fluconazole, posaconazole prophylaxis yielded even lesser fungal related mortality and significantly decreased invasive fungal infection rate. Considering the fact that posaconazole is already being used for acute myeloid leukemia (AML) and myelodysplastic syndromes patients undergoing induction treatment, it is only natural that posaconazole be used for AA/hMDS patients, who are at higher risk of developing invasive fungal infection compared to AML.

ELIGIBILITY:
Inclusion Criteria:

1. willing and able to provide written informed consent for voluntary participation in the trial
2. adult patients (≥18 years, <75 years old)
3. no QTc prolongation on initial ECG
4. Adequate organ function for treatment as follows:

A. Absolute neutrophil count > 1.5 x 109/L B. Platelets >100 x 109/L C. Serum creatinine ≤ 2.0 x ULN (upper limit of normal) D. Serum bilirubin ≤ 1.5 x ULN E. AST and ALT ≤ 2.0 x ULN

Exclusion Criteria:

1. those suspected of fungal infection within 30 days of ATG treatment
2. those allergic to -triazoles
3. those with history of malignancies within 5 years and/or concomitant malignancy other than AA/hMDS
4. those with history of chemotherapy, radiotherapy and/or other immunosuppressants
5. female patients who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
6. active HBV, HCV patients
7. HIV positive patients
8. those with history of receiving organ transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Posaconazole Prophylaxis Group: aplastic anemia / hypoplastic myelodysplastic syndrome patients undergoing antithymocyte globulin treatment and receiving posaconazole as prophylaxis antifungal agent
  Posaconazole: Dosing of posaconazole Posaconazole tablet 300 mg twice daily on day 1; Maintenance dose: 300 mg once daily on day 2 and thereafter. Treatment period: 4 weeks
  *if posaconazole tablet intolerance: posaconazole suspension 200mg tid
Period: Overall Study
Arm/Group | Posaconazole Prophylaxis Group
Started | 20
Completed | 14
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Posaconazole Prophylaxis Group
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/ Not Hispanic or Latino | 20
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 20

OUTCOME MEASURES:

1. Primary Outcome: the Incidence of Proven/Probable/Possible Fungal Infection
Description: Define Invasive fungal infections according to guidelines of the Invasive Fungal Infections Cooperative Group of the European Organization for Research and Treatment of Cancer and Mycoses Study Group of the National Institute of Allergy and Infectious Diseases (Ascioglu S, Rex JH, de Pauw B, et al. Defining opportunistic invasive fungal infections in immunocompromised patients with cancer and hematopoietic stem cell transplants: an international consensus. Clin Infect Dis. 2008;46:1813-1821.
Time Frame: during 4 weeks of posaconazole prophylaxis (i.e. upto 4 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Posaconazole Prophylaxis Group
Number analyzed (Participants) | 20
Participants | 20

2. Secondary Outcome: Overall Survival
Description: The overall survival (OS) curves will be estimated using the Kaplan-Meier method
Time Frame: through study completion, an average of 18 months
Reporting Status: Not Posted

3. Secondary Outcome: Any Incidence of Proven/Probable/Possible Fungal Infection
Description: as for outcome 1
Time Frame: through study completion, an average of 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: Definition of adverse event and serious adverse event, used to collect adverse event informations are not differs from the clinicaltrials.gov definitions.
Arm/Group | Posaconazole Prophylaxis Group
All-Cause Mortality (participants affected / at risk) | 6/20
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Posaconazole Prophylaxis Group (N=20)
Herpes zoster (Infections and infestations) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Cellulitis (Infections and infestations) | 1
Cardiac arrest (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Posaconazole Prophylaxis Group (N=20)
Liver function abnormality (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT03318159/Prot_SAP_ICF_000.pdf